CLINICAL TRIAL: NCT01414543
Title: Counselling and Clinical Psychologists Lived Experience of Client Violence
Brief Title: Psychologists' Lived Experience of Client Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East London (Other)
Responsible Party: Principal Investigator, Fardin Jussab, Dr, University of East London
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UEL1
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2009-08

CONDITIONS: Life Experiences
Keywords: violence
MeSH Terms: interventions — Consent Forms; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- providing information sheet (Other): providing participants with information regarding the purpose of the research
  Interventions: Other: Information Sheet
- Seeking consent (Other)
  Interventions: Other: Consent
- Interview Participant (Other)
  Interventions: Other: interview
- Debrief (Other): The Participants will be debriefed after the interview.
  Interventions: Other: Debrief

INTERVENTIONS:
Other: Information Sheet — Providing the Participant with information regarding the aim of the experiment
  Arms: providing information sheet
Other: Consent — Providing a consent form for participants. The participant is aware of his or her rights
  Arms: Seeking consent
Other: interview — participants will interviewed by fardin jussab for approximately one hour regarding their experience of client violence
  Arms: Interview Participant
Other: Debrief — at the end of each interview the researcher will ask participants whether the emotions aroused in the interview require further discussions. Interviewees will be also advised that should they wish to talk further about any topics covered the in the interview, they could telephone the researcher at a later time. There will also be leaflets of supporting agencies.
  Arms: Debrief

SUMMARY:
The objective of the proposed research is to gain a detailed understanding and account of psychologists' experience of client violence in clinical practice. The emphasis is upon a detailed understanding of how psychologists perceive and understand their experience of client violence and its impact upon their identity as clinicians and as individuals.

DETAILED DESCRIPTION:
This research is interested in Counselling and Clinical Psychologists who have experienced client violence at their work place. The main research question being asked is how do psychologists' understand their personal experiences of client violence. This is an important and interesting subject for Counselling and Clinical Psychologists as it provides a detailed personal account of the implications of violence upon their personal and professional identity, psychological well being and how they define violence. Furthermore, this research may help facilitate in designing a specific policy and help future research to issue guidelines for counselling and clinical psychologists in order to keep themselves safe within their professional practice. Psychologists working for the National Health Service will be recruited and provided with information regarding the research aims and objectives. There will be interviews held at their place of work for approximately one hour.

ELIGIBILITY:
Inclusion Criteria:

* Psychologist's who have experienced client violence

Exclusion Criteria:

-

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
experience of violence | one hour
  participant's discuss their experince of client violence in the work place

CONTACTS AND LOCATIONS:
Overall Officials: Helen Murphy, BA, MSc, DPhil, Study Chair — University of East London
Locations (1):
- National Health Service, London, United Kingdom